CLINICAL TRIAL: NCT04903951
Title: A Single-center, Randomized, Open Label, Parallel Arm, Prospective Study to Evaluate the Impact of Early Ventilation in Stroke Outcomes in Patients With Sleep Apnea After First Ever Stroke
Brief Title: Impact of Early Ventilation in Stroke Outcomes in Patients With Sleep Apnea After First Ever Stroke
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philips Portuguesa S.A. (Industry)
Responsible Party: Principal Investigator, Sílvia Correia, Principal Investigator, Philips Portuguesa S.A.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSASV-01-01
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Sleep Apnea
Keywords: stroke; early ventilation; sleep apnea
MeSH Terms: conditions — Stroke; Sleep Apnea Syndromes; Respiratory Aspiration | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASV therapy + best medical treatment for stroke, including rehabilitation (Experimental): Adaptive Servoventilation (ASV) therapy plus best medical treatment for stroke, including rehabilitation.
  Interventions: Device: Adaptive Servoventilation (ASV) therapy; Other: Best medical treatment
- Best medical treatment for stroke, including rehabilitation (Active Comparator): Best medical treatment for stroke, including rehabilitation.
  Interventions: Other: Best medical treatment

INTERVENTIONS:
Device: Adaptive Servoventilation (ASV) therapy — Patients assigned to the active group will receive ventilatory support with ASV (DreamStation BiPAP autoSV®) during diurnal and nocturnal sleep, from study randomization until clinically indicated
  Arms: ASV therapy + best medical treatment for stroke, including rehabilitation
Other: Best medical treatment — Best medical treatment for stroke, including rehabilitation

SUMMARY:
To evaluate the impact of early ventilation in stroke outcomes in patients with sleep apnea and first ever stroke, 1 month after stroke.

DETAILED DESCRIPTION:
Single-center, randomized, open label, parallel arm, prospective study in patients with sleep apnea after first-ever stroke.

The study will consist of screening, baseline assessment, interventional period (consisting of a treatment period and follow-up visits), and a follow-up phone call.

Patients will be randomly assigned to ASV (active) or control groups, within 4 days after the PSG II and will start the respective intervention in the same day.

Patients assigned to the active group will receive ventilatory support with ASV (DreamStation BiPAP autoSV®) during diurnal and nocturnal sleep, from study randomization until clinically indicated. Patients assigned to control group will receive best medical treatment for stroke alone, including rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the participant or the legally acceptable representative, prior to any study-related procedure.
2. Male or female between 18 and 80 years, inclusive, at the time of signing the informed consent.
3. Admission to the hospital within 48 h of stroke symptoms onset.
4. Ischemic first stroke diagnosis.
5. NIHSS ≥2 at screening.
6. Sleep apnea with AHI ≥15.

Exclusion Criteria:

1. CSA with Left Ventricular Ejection Fraction ⩽45%.
2. Ventilation treatment for sleep apnea diagnosis, prior to stroke.
3. Risk of aspiration.
4. Nasogastric feeding tube.
5. Transient ischemic attack, hemorrhagic stroke or subarachnoid hemorrhage.
6. Stroke due to a secondary cause (e.g. vascular malformation, vasculitis, brain tumor, head trauma, or predisposition to bleeding).
7. Cardiorespiratory distress.
8. Advanced chronic lung disease requiring supplemental oxygen.
9. Concomitant central nervous system diseases such as dementia or multiple sclerosis.
10. Uncontrolled psychosis or agitation.
11. Glasgow Coma Scale (GCS) score <10 at screening.
12. Anosognosia, global or Wernicke aphasia.
13. Insufficient upper limbs function to use a mask and no overnight caregiver to help.
14. Inability to attend to the rehabilitation program of the hospital.
15. Pregnant and breast-feeding women.
16. Participation in another clinical study (except a standard-of-care registry).
17. Any other condition that, according to the Investigator, renders the subject unsuitable for ventilation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with improvement in neurological parameters (reduction of ≥1 point from the beginning in Rankin scale) 1 month after stroke. | 1 month after stroke

SECONDARY OUTCOMES:
Proportion of patients with improvement in neurological parameters (reduction of ≥1 point from the beginning in Rankin scale) at 4 and 6 months after stroke. | 4 and 6 months after stroke
Change from baseline in National Institutes of Health Stroke Scale (NIHSS) to measure improvement in neurological parameters at month 1, 4 and 6 after stroke. | 1, 4 and 6 months after stroke
Type II full polysomnography (PSG II) within 7 days of stroke symptoms onset in all patients with AHI >5 as assessed by ApneaLink™ | Within 7 days after admission
Adherence in the Servoventilation group | After 1, 4 and 6 months
  % nights of device use; average hours per night of device use
Efficacy in the Servoventilation group | After 1, 4 and 6 months
  Apnea-Hypopnea Index
Adverse events monitoring | Through study completion, an average of 2 years
  All AEs occurring within the period of observation for the clinical study must be fully evaluated, documented, reported (if applicable) and archived.
Cardiovascular events evaluation at month 1, 4 and 6 months after stroke in randomized patients | 1, 4 and 6 months after stroke
Cardiovascular events evaluation 12 months after stroke in all participants. | 12 months after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Sílvia Correia, MD, Principal Investigator — Trofa Saúde Hospital
Locations (1):
- Unidade Local de Saúde de Matosinhos, Matosinhos Municipality, Portugal

IPD SHARING:
Plan to Share IPD: No